CLINICAL TRIAL: NCT01552213
Title: A Randomized Controlled Trial of Early Screening and Treatment of Women With Prediabetes in Pregnancy
Brief Title: Early Screening and Treatment of Women With Prediabetes in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Santa Clara Valley Medical Center (Other)
Responsible Party: Principal Investigator, Yasser Yehia El-Sayed, Professor of Obstetrics & Gynecology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23445
Record Dates: First submitted 2012-03-06; First posted 2012-03-13 (Estimated); Results first posted 2019-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2018-07

CONDITIONS: Diabetes; Pregnancy
MeSH Terms: conditions — Diabetes Mellitus | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment for glucose intolerance (Active Comparator): Regular visit with dietician, exercise, self blood glucose monitoring, Insulin therapy if determined necessary.
  Interventions: Other: Treatment for glucose intolerance
- Minimum intervention control group (Active Comparator): Single visit with dietician or health educator followed by routine care per provider.
  Interventions: Other: Minimum intervention control group

INTERVENTIONS:
Other: Minimum intervention control group — A single visit with a dietician or health educator to discuss general health risks, good eating habits, and appropriate weight gain. This will be followed by routine prenatal care per provider.
  Arms: Minimum intervention control group
Other: Treatment for glucose intolerance — Diet, exercise glucose monitoring, insulin if necessary
  Arms: Treatment for glucose intolerance

SUMMARY:
The investigators hope to learn whether treatment with medical nutrition therapy (MNT) for pregnant women with prediabetes decreases the rate and severity of impaired glucose tolerance later in pregnancy and improves perinatal outcomes. Given the rising rates of obesity and diabetes in this country even among young women and the adverse affects of diabetes of pregnant women and their infants, the investigators feel that it is important to not only identify women at high risk for diabetes early in pregnancy but determine the appropriate management strategy

DETAILED DESCRIPTION:
INTAKE VISIT: A health professional performs this visit soon after the diagnosis of pregnancy. Standardized glycosylated hemoglobin (A1C)is drawn as part of the routine prenatal panel at the above institutions. Women with an A1C of >6.5% are categorized as having type 2 diabetes, excluded from randomization, and referred for medical nutrition therapy, blood glucose monitoring, and insulin as needed. Women with an initial A1C <5.7% will receive routine prenatal care by their usual providers and will be screened for gestational diabetes Mellitus (GDM) in the second trimester per routine. Standard treatment for both these diabetic groups will be provided independently of this study, but anonymous outcome data will be available via hospital perinatal databases. Women with an A1c of 5.7-6.4% are eligible for the study.

EARLY PRENATAL VISIT: women with an A1C of 5.7-6.4% will be informed by their providers that they fall into a group labeled "prediabetes" outside of pregnancy and will be invited to learn about the study. All prediabetic women (agreeing to enroll or not) will be informed about general health risks and appropriate weight gain during pregnancy. Women who enroll will be queried regarding basic demographic information, pre-pregnancy weight, height, and obstetric and family history. Standardized weight, blood pressure (BP), and body mass index (BMI) will be recorded. Participants will be given a 1-page survey regarding their knowledge of risk factors for diabetes, appropriate weight gain in pregnancy, and the benefits of breastfeeding.

RANDOMIZATION AND MANAGEMENT: Women who enroll by 13 weeks gestation will be stratified by BMI < 30 or > 30 and randomized to either:

1. Minimal Intervention (Control) Group: A single visit with a randomized control trial (RCT)-associated dietitian or health educator to discuss general health risks, good eating habits, and appropriate weight gain. This will be followed by routine prenatal care as determined by provider.
2. Treatment Group: Treatment for glucose intolerance including:

Diet: Regular visits with a dietitian every 2 weeks emphasizing a food and beverage plan (Institute of Medicine standards) of appropriate energy and no more than 45% carbohydrate; limited saturated fat; adequate protein, mineral and vitamin intake; and portion control by 'carbohydrate counting'. Food and beverage intake will be divided into 3 meals and 3 snacks and self-recorded on daily food records. Recommended choices of foods and carbohydrate type will take into account personal and cultural preferences. Standardized weight will be measured and charted at each visit. The MNT plan will be adjusted according to maternal weight gain and ongoing glycemic levels. Participants will continue the MNT plan until delivery, and it will be adjusted postpartum for the needs of breastfeeding. Furthermore this group will be treated with:

A. EXERCISE: Participants will be encouraged to exercise with a minimum of brisk walking for 30 minutes each day (often 10 minutes after each meal).

B. SELF BLOOD GLUCOSE MONITORING: Participants will perform finger sticks four times each day (fasting and 1-hour after starting breakfast, lunch, and dinner) and self-recording of these values. At study visits the accuracy of the written records will be compared to the meter memory, and the glucose values will be downloaded for later analysis. The One Touch Delica and UltraMini self-monitoring of blood glucose (SMBG) system will be used and the meter, lancets and strips will be provided free of charge to the participants.

C. INSULIN: Participants will be started on insulin therapy by standard methods if more than 25% of fasting finger sticks are greater than 99 mg/dL or 1-hour post prandial finger sticks are greater than 135 mg/dL over a 2-week interval.

26 WEEKS GESTATION: Participants in both groups will be assessed for weight gain and blood pressure, and they will complete a 75-g, 2-hr oral glucose tolerance test (OGTT) (2H GTT). Those in the minimal intervention group with one or more abnormal value by ADA standards will be treated for GDM. No additional intervention will be given to women in the treatment group since will already be receiving treatment. In this study, we have chosen to use the 2H GTT as it has been correlated with adverse perinatal outcomes as described by the Hyperglycemia and Adverse Pregnancy Outcome (HAPO) study group.

DELIVERY: Recommendations for timing of delivery, management of labor, and route of delivery will be made by usual obstetric care providers independent of study personnel. All participants will have A1C measured as an indicator of late pregnancy glycemic control. Umbilical cord blood will be collected on all participants to evaluate levels of c-peptide. Elevated c-peptide is a measure of fetal hyperinsulinemia and a marker of fetopathy24. Delivery and neonatal data will be collected (see below). Participants will be instructed to continue the diet therapy for at least 6 months postpartum

6-WEEK POSTPARTUM VISIT: All participants will undergo a 2H GTT and have A1C checked. Their weight will be recorded and compared to pre-pregnancy weight. Breastfeeding will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Singleton pregnancy
* Prenatal care established at less than 14 weeks
* A1C 5.7-6.4%
* Delivery planned at Lucille Packard Children's Hospital at Stanford University (LPCH) or Santa Clara Valley Medical Center (SVMC)

Exclusion Criteria:

* preexisting diabetes or chronic steroid use
* known major fetal anomalies

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2012-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Y El-Sayed, MD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Santa Clara Valley Medical Center, San Jose, California
  - Stanford University School of Medicine/Lucile Packard Childrens Hospital, Stanford, California

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment for Glucose Intolerance | Minimum Intervention Control Group
Started (Number of subjects randomized) | 50 | 45
Analyzed (Subjects who completed the OGTT or were started on insulin prior to the OGTT) | 42 | 41
Completed (Pregnancy outcome data available) | 37 | 37
Not Completed | 13 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment for Glucose Intolerance | Minimum Intervention Control Group | Total
Number analyzed (Participants) | 42 | 41 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.4 (5.1) | 34.3 (5.2) | 33.4 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 41 | 83
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With a Diagnosis of Gestational Diabetes at 26 Weeks Gestation.
Description: Diagnosis based on criteria recommended by the ADA (Oral GTT with one abnormal value, fasting greater than or equal to 92, on hour greater than or equal to 180, two hour greater than or equal to 153)
Time Frame: 26 weeks of gestation
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment for Glucose Intolerance | Minimum Intervention Control Group
Number analyzed (Participants) | 42 | 41
Participants | 19 | 23
Statistical Analysis 1: Comparison: Treatment for Glucose Intolerance vs Minimum Intervention Control Group; Test type: Superiority; p = 0.32, Chi-squared; Risk Ratio (RR) = 0.80, 95% CI 2-sided [0.53 to 1.24]

2. Secondary Outcome: Number of Participants With Different Modes of Delivery
Description: Modes of delivery investigated were: cesarean delivery, vaginal delivery, assisted vaginal delivery, spontaneous delivery and termination of pregnancy.
Time Frame: Duration of pregnancy. Pregnancy expected to last up to 40 weeks gestation
Population: Participants with available data included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment for Glucose Intolerance | Minimum Intervention Control Group
Number analyzed (Participants) | 40 | 38
Participants
  Cesarian delivery | 11 | 17
  Vaginal delivery | 26 | 19
  Assisted vaginal | 0 | 1
  Spontaneous abortion | 2 | 1
  Termination | 1 | 0
Statistical Analysis 1: Comparison: Treatment for Glucose Intolerance vs Minimum Intervention Control Group; Test type: Superiority; p = 0.32, Chi-squared

3. Secondary Outcome: Number of Participants With Excessive Gestational Weight Gain
Description: Excessive weight gain greater than the Institute of Medicine guidelines
Time Frame: Duration of pregnancy. Pregnancy expected to last up to 40 weeks gestation
Population: Participants with available data included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment for Glucose Intolerance | Minimum Intervention Control Group
Number analyzed (Participants) | 35 | 36
Participants | 6 | 6
Statistical Analysis 1: Comparison: Treatment for Glucose Intolerance vs Minimum Intervention Control Group; Test type: Superiority; p = 0.96, Chi-squared

4. Secondary Outcome: Mean Hemoglobin A1C Value at Delivery
Time Frame: Duration of pregnancy. Pregnancy expected to last up to 40 weeks gestation
Population: Participants with available data included in the analysis.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Treatment for Glucose Intolerance | Minimum Intervention Control Group
Number analyzed (Participants) | 28 | 28
percent | 5.5 (0.3) | 5.8 (0.4)
Statistical Analysis 1: Comparison: Treatment for Glucose Intolerance vs Minimum Intervention Control Group; Test type: Superiority; p = 0.01, t-test, 2 sided

5. Secondary Outcome: Mean Fasting Triglyceride Level
Time Frame: Duration of pregnancy. Pregnancy expected to last up to 40 weeks gestation
Population: Participants with available data included in the analysis.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment for Glucose Intolerance | Minimum Intervention Control Group
Number analyzed (Participants) | 40 | 38
mg/dL | 181 (66.0) | 177.5 (51.5)
Statistical Analysis 1: Comparison: Treatment for Glucose Intolerance vs Minimum Intervention Control Group; Test type: Superiority; p = 0.75, t-test, 2 sided

6. Secondary Outcome: Number of Patients With Gestational Hypertension
Description: Hypertensive disorder in pregnancy with blood pressure greater than or equal to 140/90 after 20 weeks gestation
Time Frame: Duration of pregnancy. Pregnancy expected to last up to 40 weeks gestation
Population: Participants with available data included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment for Glucose Intolerance | Minimum Intervention Control Group
Number analyzed (Participants) | 38 | 36
Participants | 3 | 3
Statistical Analysis 1: Comparison: Treatment for Glucose Intolerance vs Minimum Intervention Control Group; Test type: Superiority; p = 0.95, Chi-squared

7. Secondary Outcome: Number of Patients With Pre-eclampsia
Description: Blood pressure greater than or equal to 140/90 with 300 mg of protein on a 24-hour urine collection.
Time Frame: Up to 6 weeks after delivery
Population: Participants with available data included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment for Glucose Intolerance | Minimum Intervention Control Group
Number analyzed (Participants) | 50 | 45
Participants | 2 | 2
Statistical Analysis 1: Comparison: Treatment for Glucose Intolerance vs Minimum Intervention Control Group; Test type: Superiority; p = 0.5, Chi-squared

8. Secondary Outcome: Mean Level of Postpartum Oral Glucose-tolerance-test at 6 Weeks Postpartum
Time Frame: 6 weeks after delivery
Population: Participants with available data included in the analysis.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment for Glucose Intolerance | Minimum Intervention Control Group
Number analyzed (Participants) | 23 | 28
mg/dL | 115.8 (46.5) | 108.9 (41.1)
Statistical Analysis 1: Comparison: Treatment for Glucose Intolerance vs Minimum Intervention Control Group; Test type: Superiority; p = 0.6, t-test, 2 sided

9. Secondary Outcome: Number of Participants With Need for Insulin Therapy
Description: Insulin required during pregnancy
Time Frame: Duration of pregnancy. Pregnancy expected to last up to 40 weeks gestation
Population: Participants with available data included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment for Glucose Intolerance | Minimum Intervention Control Group
Number analyzed (Participants) | 39 | 38
Participants | 14 | 10
Statistical Analysis 1: Comparison: Treatment for Glucose Intolerance vs Minimum Intervention Control Group; Test type: Superiority; p = 0.36, Chi-squared

10. Secondary Outcome: Mean Neonatal Birth Weight
Time Frame: Duration of pregnancy. Pregnancy expected to last up to 40 weeks gestation
Population: Participants with available data included in the analysis.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Treatment for Glucose Intolerance | Minimum Intervention Control Group
Number analyzed (Participants) | 42 | 41
grams | 3218 (611) | 3322 (473)
Statistical Analysis 1: Comparison: Treatment for Glucose Intolerance vs Minimum Intervention Control Group; Test type: Superiority; p = 0.42, t-test, 2 sided

11. Secondary Outcome: Mean Ponderal Index
Description: The Corpulence Index (CI) or Ponderal Index (PI) is a measure of leanness (corpulence) of a person calculated as a relationship between mass and height.
Time Frame: Duration of pregnancy. Pregnancy expected to last up to 40 weeks gestation
Population: Participants with available data included in the analysis.
Measure: Mean (Standard Deviation); unit: kg/m3
Arm/Group | Treatment for Glucose Intolerance | Minimum Intervention Control Group
Number analyzed (Participants) | 36 | 36
kg/m3 | 2.5 (0.3) | 2.5 (0.3)
Statistical Analysis 1: Comparison: Treatment for Glucose Intolerance vs Minimum Intervention Control Group; Test type: Superiority; p = 0.5, t-test, 2 sided

12. Secondary Outcome: Mean Level of Umbilical Cord C-peptide >=90th Percentile in the Whole Cohort
Description: C-peptide test is a tool for monitoring and treating diabetes.
Time Frame: Duration of pregnancy. Pregnancy expected to last up to 40 weeks gestation
Population: Participants with available data included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment for Glucose Intolerance | Minimum Intervention Control Group
Number analyzed (Participants) | 23 | 17
Participants | 3 | 1
Statistical Analysis 1: Comparison: Treatment for Glucose Intolerance vs Minimum Intervention Control Group; Test type: Superiority; p = 0.46, Chi-squared

13. Secondary Outcome: Number of Participants With Neonatal Hypoglycemia
Description: Infants treated for neonatal hypoglycemia-- Glucose of <36 mg/dl; <2 millimoles (mM)
Time Frame: 1 week after delivery
Population: Participants with available data included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment for Glucose Intolerance | Minimum Intervention Control Group
Number analyzed (Participants) | 35 | 36
Participants | 2 | 2
Statistical Analysis 1: Comparison: Treatment for Glucose Intolerance vs Minimum Intervention Control Group; Test type: Superiority; p = 1, Chi-squared

14. Secondary Outcome: Number of Participants With Neonatal Hyperbilirubinemia
Description: Neonates treated for hyperbilirubinemia
Time Frame: 1 week after delivery
Population: Participants with available data included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment for Glucose Intolerance | Minimum Intervention Control Group
Number analyzed (Participants) | 36 | 36
Participants | 9 | 6
Statistical Analysis 1: Comparison: Treatment for Glucose Intolerance vs Minimum Intervention Control Group; Test type: Superiority; p = 0.56, Chi-squared

15. Secondary Outcome: Number of Participants With Intrauterine Fetal Demise
Time Frame: Duration of pregnancy and up to 28 days after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment for Glucose Intolerance | Minimum Intervention Control Group
Number analyzed (Participants) | 37 | 37
Participants | 0 | 1

ADVERSE EVENTS:
Arm/Group | Treatment for Glucose Intolerance | Minimum Intervention Control Group
Serious Adverse Events (participants affected / at risk) | 0/50 | 1/45
Other Adverse Events (participants affected / at risk) | 0/50 | 0/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment for Glucose Intolerance (N=50) | Minimum Intervention Control Group (N=45)
Intrauterine Fetal Demise (Pregnancy, puerperium and perinatal conditions) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No